CLINICAL TRIAL: NCT04886232
Title: A Prospective, Multicenter, Randomized, Comparator-controlled, Evaluator-blinded Study to Evaluate the Safety and Effectiveness of VP1 Lido US for Volume Augmentation of the Cheek
Acronym: BCheek
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M930061001
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cheek Volume Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VP1 Lido US - NC (Experimental): Injection to the left cheek via needle and to the right cheek via canula
  Interventions: Device: VP1 Lido US
- VP1 Lido US - CN (Experimental): Injection to the left cheek via canula and to the right cheek via needle
  Interventions: Device: VP1 Lido US
- Restylane Lyft Lidocaine - NC (Active Comparator): Injection to the left cheek via needle and to the right cheek via canula
  Interventions: Device: Restylane Lyft Lidocaine
- Restylane Lyft Lidocaine - CN (Active Comparator): Injection to the left cheek via canula and to the right cheek via needle
  Interventions: Device: Restylane Lyft Lidocaine

INTERVENTIONS:
Device: VP1 Lido US — Hyaluronic acid dermal filler containing lidocaine
  Arms: VP1 Lido US - CN; VP1 Lido US - NC
Device: Restylane Lyft Lidocaine — Hyaluronic acid dermal filler containing lidocaine
  Arms: Restylane Lyft Lidocaine - CN; Restylane Lyft Lidocaine - NC

SUMMARY:
The primary objective of the study is to demonstrate non-inferiority of VP1 Lido US versus an approved hyaluronic acid dermal filler following deep (subdermal and/or supraperiosteal) injection of the cheek for volume augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Has a symmetrical rating of 2 (moderate) or 3 (severe) for right and left cheek on the Merz Cheeks Fullness Assessment Scale (MCFAS)
* Desires cheek augmentation to correct volume deficit in the midface and is willing to receive sufficient volume to achieve at least a 1-point improvement on the MCFAS

Exclusion Criteria:

* Skin or fat atrophy in the midfacial region other than that related to age.
* Subjects with body mass index of <18.5 or ≥30
* Acute inflammatory process or active infection at the injection site (e.g., acne, eczema, streptococcus infections), or history of chronic or recurrent infection or inflammation with the potential to interfere with the study results or increase the risk of AEs.
* Prior surgery, including midfacial plastic surgery, or has a permanent implant or graft in the midfacial region that could interfere with effectiveness assessments.
* Received midfacial region treatments with porcine-based collagen fillers or with RADIESSE® or with volumizing hyaluronic acid fillers such as but not limited to Juvéderm® Voluma, Restylane® Lyft within the past 24 months and/or with other HA fillers or mesotherapy within the past 12 months or plans to receive such treatments during participation in the study.
* Received facial dermal therapies (i.e., facial ablative or fractional laser, dermabrasion, chemical peels, non-invasive skin-tightening [e.g., Ultherapy®, Thermage®] and surgical procedures) in the midfacial region within the past 12 months or plans to receive them in the facial region during participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 12 on the Merz Cheeks Fullness Assessment Scale (MCFAS) | Baseline to week 12
  The MCFAS is a 5-point ordinal rating

SECONDARY OUTCOMES:
Change from baseline to Week 12 on the MCFAS by injection type (cannula, needle) | Baseline to week 12
Treatment response rate where response is defined as a ≥ 1-point improvement on both cheeks when comparing the change from baseline to Week 12 | Baseline to week 12
FACE-Q satisfaction with cheeks for treated subjects at baseline and Week 12 | Week 12
Global Aesthetic Improvement Scale (GAIS) scores for treated subjects at Week 12, as completed by the treating investigator | Week 12
GAIS scores for treated subjects at Week 12, as completed by the subject | Week 12
Responder rates at Week 12, according to the MCFAS, as assessed by three blinded board-certified Independent Panel Reviewers (IPRs) using subject photographs | Week 12
Incidence of related serious or delayed onset adverse events (>21 days after treatment) following the first treatment including touch-up until Week 48 | Baseline to week 48

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (10):
- Germany (10):
  - Hautmedizin Bad Soden, Merz Investigational Site #0490189, Bad Soden am Taunus
  - Rosenparkklinik, Merz Investigational Site #0490099, Darmstadt
  - Praxis für Hautkrankheiten, Merz Investigational Site #0490375, Drensteinfurt
  - Dermatologic Private Practive, Merz Investigational Site #0490381, Düsseldorf
  - Universität Hamburg, Merz Investigational Site #0490095, Hamburg
  - Dermatologic Private Practice, Merz Investigational Site #0490345, Hamburg
  - Private Clinic, Merz Investigational Site #0490284, Mannheim
  - Privatpraxis für Dermatologie und Ästhetik, Merz Investigational Site #0490371, München
  - Haut- und Lasercentrum Potsdam, Merz Investigational Site #0490362, Potsdam
  - Centroderm GmbH, Merz Investigational Site #0490367, Wuppertal

IPD SHARING:
Plan to Share IPD: No